CLINICAL TRIAL: NCT06189170
Title: A Phase I, Randomised, Double-Blinded, Placebo-Controlled Study to Evaluate KP405. Part 1: Single Ascending Dosing in Healthy Participants. Part 2: Multiple Ascending Dosing in Healthy Participants and Parkinson's Disease Patients.
Brief Title: Phase I Study to Evaluate KP405 in Healthy and Parkinson's Disease Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kariya Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KP405CS01
Record Dates: First submitted 2023-11-13; First posted 2024-01-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Safety Issues; Tolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Cohort 1 (Experimental): KP405_dose 1, single dose
  Interventions: Drug: KP405; Drug: Placebo
- Cohort 2 (Experimental): KP405_dose 2, single dose
  Interventions: Drug: KP405; Drug: Placebo
- Cohort 3 (Experimental): KP405_dose 3, single dose
  Interventions: Drug: KP405; Drug: Placebo
- Cohort 4 (Experimental): KP405_dose 4, single dose
  Interventions: Drug: KP405; Drug: Placebo
- Cohort 5 (Experimental): KP405_dose 5, single dose
  Interventions: Drug: KP405; Drug: Placebo
- Cohort 6 (Experimental): KP405_dose 6, single dose
  Interventions: Drug: KP405; Drug: Placebo
- Cohort 7 (Experimental): KP405_dose 1, multiple dose
  Interventions: Drug: KP405; Drug: Placebo
- Cohort 8 (Experimental): KP405_dose 2, multiple dose
  Interventions: Drug: KP405; Drug: Placebo
- Cohort 9 (Experimental): KP405_dose 3, multiple dose
  Interventions: Drug: KP405; Drug: Placebo
- Cohort 10 (Experimental): KP405_dose 4, multiple dose
  Interventions: Drug: KP405; Drug: Placebo
- Cohort 11 (Experimental): KP405_dose 5, multiple dose
  Interventions: Drug: KP405; Drug: Placebo

INTERVENTIONS:
Drug: KP405 — Experimental drug
Drug: Placebo — Placebo

SUMMARY:
This study will explore the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of KP405 as a potential new treatment for Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on medical evaluation including medical history, physical examination, concomitant medication, vital signs, 12-lead ECG, cardiac Holter monitoring and clinical laboratory evaluations.
* Clinical diagnosis of Parkinson's disease meeting United Kingdom Brain Bank criteria.

Exclusion Criteria:

* Clinically relevant history of abnormal physical or mental health interfering with the study as determined by medical history and physical examinations obtained during Screening as judged by the Investigator (including [but not limited to], neurological, psychiatric, endocrine, cardiovascular, respiratory, gastrointestinal, hepatic, or renal disorder), excluding Parkinson's disease.
* Clinically significant, as judged by the Investigator, neurologic disorder (other than Parkinson's disease) including history of stroke or transient ischaemic attack within 12 months of Screening, cognitive impairment, seizure within 5 years of Screening or head trauma with loss of consciousness within 6 months of Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse event (AE) reporting | Through study completion, an average of 1 year
  Clinical safety data from adverse event (AE) reporting
12-lead electrocardiogram (ECG) | Through study completion, an average of 1 year
  Clinical safety data from 12-lead electrocardiogram (ECG) machine will automatically calculate:
  RR interval PR interval QRS complex QT interval QTcF (QT interval corrected for heart rate using Fridericia's formula) Heart rate (beats per minute)
Continous ECG monitoring | Through study completion, an average of 1 year
  Clinical safety data from cardiac Holter monitoring
Blood pressure | Through study completion, an average of 1 year
  Clinical safety data from supine blood pressure (mmHg)
Pulse rate | Through study completion, an average of 1 year
  Clinical safety data from pulse rate (beats per minute)
Temperature | Through study completion, an average of 1 year
  Clinical safety data from oral temperature (degrees Celcius)
Biochemistry parameters in blood samples | Through study completion, an average of 1 year
  Blood chemistry clinical safety data from blood samples. The measurements are:
  Amylase BUN Creatinine Glucose Sodium Potassium Phosphate Chloride Calcium AST ALT GGT Alkaline phosphatase Total bilirubin Uric acid Albumin Total protein Lactate dehydrogenase
Haematology parameters in blood samples | Through study completion, an average of 1 year
  Haematology clinical safety data from blood samples. The measurements are:
  Haemoglobin Haematocrit RBC count RBC indices (MCV, MCH, MCHC) Platelet count White blood cell count with differential
Urine samples | Through study completion, an average of 1 year
  Clinical safety data from urinalysis (dipstick*). The following will be measured:
  Glucose Bilirubin Ketone Specific Gravity Blood pH Protein Urobilinogen Nitrite Leukocyte Esterase
  *Microscopic analysis if dipstick is abnormal
  Drugs of abuse:
  Amphetamines Barbiturates Benzodiazepines Cocaine Cannabinoids Opiates
Coagulation parameters in blood samples | Through study completion, an average of 1 year
  Coagulation clinical safety data from blood samples. The measurements are:
  Prothrombin time International normalisation ratio Activated partial thromboplastin time
Serology parameters in blood samples | Through study completion, an average of 1 year
  Serology clinical safety data from blood samples. The measurements are:
  Anti-HIV I/II Anti-HCV HBsAg
Alcohol breath test | Through study completion, an average of 1 year
  Alcohol measurements will be done as a breath test
Height | Through study completion, an average of 1 year
  As part of a full physical examination the height of the subjects will be measured (in meters)
Body weight | Through study completion, an average of 1 year
  As part of a full physical examination body weight of the subjects will be measured (in kilograms)
Assessments of body parts | Through study completion, an average of 1 year
  As part of a full physical examination assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular system, abdomen (liver and spleen), lymph nodes and extremities will be conducted
Injection site reactions | Through study completion, an average of 1 year
  Clinical safety data from injection site reactions

SECONDARY OUTCOMES:
Pharmacokinetics parameters - Cmax | 0-48 hours
  Plasma PK concentrations including but not limited to: maximum plasma concentration (Cmax) (ng/ml)
Pharmacokinetics parameters - tmax | 0-48 hours
  Plasma PK concentrations including but not limited to: time to reach Cmax (tmax) (minutes)
Pharmacokinetics parameters - AUC0-t | 0-48 hours
  Plasma PK concentrations including but not limited to: area under the plasma concentration-time curve (AUC) from zero to the last quantifiable concentration () (ng/ml x hours)
Pharmacokinetics parameters - AUC0-∞ | 0-48 hours
  Plasma PK concentrations including but not limited to: AUC from zero to infinity (AUC0-∞)(ng/ml x hours)
Pharmacokinetics parameters - AUC0-24h | 0-48 hours
  Plasma PK concentrations including but not limited to: AUC from zero to 24 hours () (ng/ml x hours)
Pharmacokinetics parameters - AUC0-48h | 0-48 hours
  Plasma PK concentrations including but not limited to: AUC from zero to 48 hours (AUC0-48h) (ng/ml x hours)
Pharmacokinetics parameters - half life | 0-48 hours
  Plasma PK concentrations including but not limited to: half life (t1/2) (hours)
Pharmacodynamic parameters-Pupillometry | Through study completion, an average of 1 year
  The pupillometry measurements will be completed in a room where ambient noise and lighting will be controlled and uniform. After resting for 5 minutes, and before and after receiving the study drug, the pupillometry measurements (repeated once) will be taken from each eye using a pupilometer with an opaque rubber cup covering one eye. Each pupillometry session measuring both eyes will be approximately 1 minute.
Pharmacodynamic parameters - EEG | Through study completion, an average of 1 year
  Absolute and relative power spectral densities (PSDs) calculated for each 1 second epoch (1-59 Hz bins). Also grouped into the standard EEG bandwidths: delta, theta, alpha, beta and gamma. Additionally, the PSD variables will be averaged across brain regions of interest, including frontal, central, parietal, temporal and occipital
Pharmacodynamic parameters - Food VAS | Through study completion, an average of 1 year
  The following questions will be asked:
  1. How hungry do you feel (from 'not hungry at all' to 'very hungry')?
  2. How full do you feel (from 'not full at all' to 'very full')?
  3. How satisfied do you feel (from 'completely empty' to 'I cannot eat more')?
  4. How much do you think you can eat now (from 'nothing at all' to 'a lot')?
Pharmacodynamic parameters- Daily Food Diary | Through study completion, an average of 1 year
  "You are required to keep an up-to-date food diary for the next few days, recording everything you consume (all nutrition that passes your lips)"
Pharmacodynamic parameters - Test Meal | Through study completion, an average of 1 year
  The test meal model is an accepted experimental method for assessing the effects of an intervention on food intake in a laboratory setting.
  In its simplest form, it involves offering participants an excess amount of pre-weighed food (a pasta-based meal), instructing participants to eat the test meal until they feel comfortably full, and then weighing the amount of food remaining once the participant has finished eating.13 The weight of food consumed can then be determined (±0.1 g) and from the nutritional information on the food packaging, energy intake (kJ) can be calculated.
Pharmacodynamic parameters - Appetite and Palatability Questionnaire | Through study completion, an average of 1 year
  This questionnaire consists of thirteen VAS questions and one multiple choice question which in sum examine the palatability of the test meal, the participants' motivation to eat, the general wellbeing and physiological sensations of the participants, and the reason why they stopped eating. The VAS questions are self-rated by the participant by putting a perpendicular marking on each of the thirteen 100 mm lines

CONTACTS AND LOCATIONS:
Overall Officials: Ezanul A Wahab, MD, Principal Investigator — MAC
Locations (1):
- MAC, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No